CLINICAL TRIAL: NCT06803472
Title: Pulsed High Intensity Laser Versus Extracorporeal Shockwave Therapy on Hypertrophic Scar Post Burn
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Fayed Ali Ibrahim, physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004524
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Hypertrophic Scar
Keywords: Hypertrophic scar
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Group A (30 patients receive pulsed high intensity laser plus taditional PT treatment for postburn hypertrophic scar.
  Groyp B (30 patients recaive extracorporeal shockwave therapy plus traditional PT treatment for post burn hypertrophic scar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group receives pulsed high intensity laser and coservative treatment (Active Comparator)
  Interventions: Device: pulsed high intensity laser therapy
- study group receives extracorporeal shockwave therapy and coservative treatment (Active Comparator)
  Interventions: Device: Extracorporeal shockwave therapy

INTERVENTIONS:
Device: pulsed high intensity laser therapy — The high-intensity laser therapy (HILT), which involves laser radiation with high-intensity, is a kind of novel and powerful . The HILT possesses its own photomechanical, photothermal, and the photo-chemical properties.
  Arms: study group receives pulsed high intensity laser and coservative treatment
Device: Extracorporeal shockwave therapy — Extracorporeal shockwave therapy is an acoustic wave that mechanically disrupts tissue by cavitation.Shock waves develop microscopic injuries in scar tissue and break down collagen fibers which lead to scar remodelin .The patient is positioned in a comfortable position. The scar site is prepared with contact gel to conduct the shock waves, 30-50 shocks/cm2 , with an energy flux density of 0.25mJ/mm2 and a frequency of 6Hz. Each treatment region is covered with 2500 to 3000 impulses with an average session time of 10-15min .
  Arms: study group receives extracorporeal shockwave therapy and coservative treatment

SUMMARY:
The goal of this clinical trial stydy : is to compare between the effect of pulsed high intensity laser and extracorporeal shockwave therapy on hypertrophic scar on post burned patients.

The main questions is it aims to answer is :

* Which is more effective on hypertrophic scar post burn Extracorporeal shockwave therapy or pulsed high intensity laser therapy?
* Participants will receive the treatment for 6 weeks.
* Assesment will be don before and after treatment.

DETAILED DESCRIPTION:
1. Subjects :

   Sixty patients have hypertrophic scar post burn. They will be selected from El Gamaa hospital and randomly distributed into two equal groups. Their ages will be ranged from 20 to 45 years.
2. Design of the study :

In this study, the patients will be randomly divided into two equal groups in number (30 patients each).

1. Group A (pulsed high intensity laser group):

   In this group of the study, thirty patients whom have hypertrophic scar post burn injury will receive pulsed high intensity laser in addition to traditional physiotherapy (deep friction massage and stretching exercises) for six weeks. The application will be three times per week.
2. Group B (Extracorporeal shockwave group):

In this group of the study, thirty patients whom have hypertrophic scar post burn injury will receive Extracorporeal shockwave therapy in addition to traditional physiotherapy (deep friction massage and stretching exercises) for six weeks. The application will be two times per week.

Equipments :

.Measurement equipments :

1. Modified Vancouver burn Scar assessment scale :

   Modified Vancouver scar scale (VSS), an observer-dependent scale of the macroscopic appearance of scarring, was used to measure changes in the scar over the period of treatment.

   The Modified Vancouver Scar Scale score is probably the most widely known scar scale that consists of three components (vascularization, pliability and scar height); the total score ranges from 0 to 11, with 0 representing normal skin.To assess 3 variables of scar characteristics: Vascularity, pliability and height.

   Scoring; vascularity ranged from 0 to 3 (1 Pink, 2 Red, 3 Purple), pliability ranged from 0 to 5 (1 Supple, 2 Yielding, 3 Firm, 4 Ropes, 5 Contracture) and height ranged from 0 to 3 (1 Less than 2 mm, 2 From 2 to 5 mm, 3 More than 5 mm). The larger the total score, the worse the HTS. The investigators choose an algebraic value for any of these characteristics based on a comparison with normal skin (zero score)
2. A Schiotz tonometer scale :

This scale will be used as an objective scale to asses the hypertrophic scar pliability and elasticity.

The tissue tonometer provides a repeatable and objective index of burn scar pliability. it is a simple, clinically useful technique for monitoring an individual's scar.

To assess scar pliability and elasticity improvement by an objective manner It is held vertically at a measured point of the scar, so the plunger moved downwards by gravity and indent the scar tissue. The instrument gives a reading on a horizontal scale numbered arbitrarily from 0 to 20, but the device does not measure scar pressure directly, a conversion table, supplied with the Schiotz tonometer pressure directly, a conversion table, supplied with the Schiotz tonometer, is used to translate the instrument readings into measurements by mmHg .

Treatment procedure :

1. Pulsed High Intensity Laser application procedure:

   * Should wear laser-protective glasses or goggles.
   * Inappropriate use of the goggles is more dangerous than their non-use, as they may provide a false sense of security.
   * Laser equipment should be placed in a controlled area with minimal access to avoid inadvertent exposure.
   * Avoid laser reflection from mirrored surfaces.
   * Avoid exposure of eyes, unclosed fontanels of children.
   * Applied at at fluence of 40 J/cm2 , pulse duration of 0.3 m/s , spot size of 5 mm in a focused mode for 3 passes.
2. Extracorporeal shockwave application procedure:

   * Patients will receive sessions of ESWT twice a week for 6 weeks.
   * ESWT will be administered on an outpatient basis; the selected treatment area is usually the most uncomfortable for the patient. Patient placed into comfortable position that allowed the vision of the treated area.
   * Each treatment region covered with 2500 to 3000 impulses with average session time 10-15 min.

conservative treatment for both groups: (Stretching exercises and Deep friction massage ) 2 sessions per week for 6 weeks

ELIGIBILITY:
Inclusion Criteria:

* The patients age will range from 20 to 45 years.
* All patients will be free from any other pathological conditions or histories except hypertrophic scar.
* patients will be selected from both gender.
* All patients will have hypertrophic scars post burn injuries.

Exclusion Criteria:

* The patients who have open wound at or near treatment site.
* The patients who have cardiac pacemakers or other implanted electronic devices.
* The patients who have any significant health problem such as diabetes, circulatory
* disorders or history of skin malignancy in the treated area.
* uncooperative patients.
* The patients who have a deep venous thrombosis (DVT).

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-26 (Estimated); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Modified Vancouver burn Scar assessment scale | change of the total score from the begginning of the treatment to the end of the treatment (after 6 weeks from the begginning of the treatment)
  Modified Vancouver scar scale , an observer-dependent scale of the macroscopic appearance of scarring, is used to measure changes in the scar over the period of treatment,The Modified Vancouver Scar Scale score is probably the most widely known scar scale that consists of three components (vascularization, pliability and scar height); the total score ranges from 0 to 11, with 0 representing normal skin ,Scoring; vascularity ranged from 0 to 3 (1 Pink, 2 Red, 3 Purple), pliability ranged from 0 to 5 (1 Supple, 2 Yielding, 3 Firm, 4 Ropes, 5 Contracture) and height ranged from 0 to 3 (1 Less than 2 mm, 2 From 2 to 5 mm, 3 More than 5 mm). The larger the total score, the worse the HTS. The investigators choose an algebraic value for any of these characteristics based on a comparison with normal skin (zero score).

SECONDARY OUTCOMES:
Aschiotz tonometer device | change of the hypertrohic scar pressure score from the begginning of the treatment to the end of the treatment (after 6 weeks from the begginning of the treatment)
  Aschiotz tonometer device, will be used as an objective scale to asses the hypertrophic scar pliability and elasticity.
  The tissue tonometer provides a repeatable and objective index of burn scar pliability. it is a simple, clinically useful technique for monitoring an individual's scar It is held vertically at a measured point of the scar, so the plunger moved downwards by gravity and indent the scar tissue. The instrument gives a reading on a horizontal scale numbered arbitrarily from 0 to 20, but the device does not measure scar pressure directly, a conversion table, supplied with the Schiotz tonometer, is used to translate the instrument readings into measurements by mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Haidy Nady Ashem, professor, Study Director — faculty of physical therapy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruchiatan K, Suhada KU, Hindritiani R, Puspitosari D, Septrina R. Combination of 1064 nm Long-Pulsed and Q-Switched Nd:YAG Laser for Facial Hypertrophic Scar and Hyperpigmentation Following Burn Injury. Int Med Case Rep J. 2022 Jan 25;15:23-27. doi: 10.2147/IMCRJ.S348091. eCollection 2022. PMID 35115845
- [Background] Lee SY, Joo SY, Cho YS, Hur GY, Seo CH. Effect of extracorporeal shock wave therapy for burn scar regeneration: A prospective, randomized, double-blinded study. Burns. 2021 Jun;47(4):821-827. doi: 10.1016/j.burns.2020.08.009. Epub 2020 Aug 29. PMID 32917473
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35115845/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32917473/